CLINICAL TRIAL: NCT00400088
Title: A Randomized, Double-blind, Double-dummy, Controlled Trial of Lithium Versus Paroxetine in Subjects With Major Depression Who Have a Family History of Bipolar Disorder or Completed Suicide - a Pilot Study
Brief Title: Lithium Versus Paroxetine in Patients With Major Depression Who Have a Family History of Bipolar Disorder or Suicide
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Julie Garnham, Dr. Claire O'Donovan, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDHA012; CDHA-RS/2006-076
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression; Bipolar Disorder; Manic Depressive Illness; Randomized Trial; Antidepressant Treatment; Lithium Treatment
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Bipolar Disorder | interventions — Paroxetine; Lithium; Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- lithium group (Experimental): Start at 600 mg po hs. Dose titrated up to a serum level of between 0.6 and 1.1 mmol/l.
  Interventions: Drug: lithium
- paroxetine group (Active Comparator): Start dose at 20 mg po od. If no clinical improvement(<20% reduction in MADRS score) by week 4 dose to be increased to 40 mg po od.
  Interventions: Drug: paroxetine

INTERVENTIONS:
Drug: paroxetine — Start at 20 mg po od. Increase dose to 40 mg po od at week 4 if there is less than 20 % reduction in MADRS scores.
  Other Names: paxil
  Arms: paroxetine group
Drug: lithium — start at 600mg po hs with dose to be flexibly titrated to a serum level of between 0.6 and 1.1 mmol/l.
  Other Names: lithane; lithium carbonate
  Arms: lithium group

SUMMARY:
This study is being done to look at how well people respond to two very different drug treatments for depression. Clinically, people with depression can respond differently to drug treatments for reasons which are not always clear. Some of our own recent research suggests that people with depression who have a family history of bipolar disorder or completed suicide, may react differently to standard antidepressant medications than those without such a family history. Our data shows that family history of completed suicide, as well as the known predictor of family history of bipolar disorder, may help identify a pre-bipolar high risk group i.e. they currently have depression but at some future date will declare a bipolar illness (manic-depression) by virtue of development of a manic episode also. Our research suggests that treatment- emergent symptoms in response to a trial of antidepressant, such as agitation may be strong predictors of future bipolarity and inherently dangerous particularly as they are not ascribed to the antidepressant treatment. Finally, it is possible that this subgroup of those with depressive illness may respond better and more safely to lithium, a mood stabiliser used in known bipolar depression.

The objective of this proposal is to investigate response to acute lithium treatment in subjects who meet the diagnostic criteria for major depression, but who are potentially at risk for bipolar disorder, by virtue of family history of bipolarity or completed suicide.

DETAILED DESCRIPTION:
Introduction: Bipolar disorder is an illness that consists of distinct episodes or "poles" of both major depression and mania (bipolar I) or major depression and hypomania (bipolar II). Both poles of the illness may be fully present simultaneously in what is referred to as a "Mixed episode". The "poles" of Major depression, Mania and Mixed mood are currently defined by descriptive criteria in the psychiatric diagnostic manual, DSMIV.

Estimates of the prevalence of Bipolar disorder are as high as 6% of the population.(1) It is a severe and potentially lethal illness which has a different course and treatment profile to unipolar depression, commonly known simply as "major depression". In 50-60% of cases however, the initial presentation of bipolar disorder is one of major depression, and several episodes of depression may occur before declaration of bipolarity, by virtue of a manic or hypomanic episode (pre-bipolar depression).(2,3) The mainstay of treatment for unipolar major depression is antidepressants. In contrast, antidepressant monotherapy is contraindicated in Bipolar I depression and must be used very cautiously in Bipolar II illness (4) with much concern for an "unacceptable cost /benefit ratio' because of the risk of antidepressant induction of mania and rapid cycling (increase in frequency of episodes as a consequence of antidepressants). (5). Hence treatment of the early depressive episodes of bipolar illness requires recognition of depression specific to bipolar disorder and appropriate choice of medication.

Unfortunately, efforts to clearly distinguish bipolar from unipolar depression cross-sectionally have been mostly disappointing. Most evidence supports the value of family history(6) and there is variable predictive value for specific phenomenological and course descriptors such as hypersomnia, psychomotor retardation, early-onset and psychotic sub types(7,8).

The dilemma then is two-fold:

1. Identifying patients suffering from major depression who are at high risk of bipolar disorder.
2. Choosing appropriate pharmacological treatment.

In choosing pharmacological treatment for a "high risk" group, there is the possibility of causing harm with antidepressants if the true diagnosis is bipolar disorder, and of not treating the depression adequately if using mood stabilizers in what is truly a unipolar illness. This dilemma applies to a large subgroup of those presenting with depression. A recent study in a primary care setting suggested that as many as 21% of patients currently treated with antidepressants for a presumed depressive disorder may in fact have a bipolar diathesis, thus representing a large group that may be improperly treated(9).

The concerns with the use of antidepressants in known bipolar depression have focused on antidepressant - induction of mania, and rapid cycling but these do not always present themselves immediately. However, there may be other subtle and immediate antidepressant treatment effects that make the diagnostic distinction possible and more pressing.(5,10)Indeed, it has been postulated that undetected bipolar depression may explain the apparent poor treatment response and increase in suicidality with the use of antidepressants in the adolescent population, where one might expect an increased prevalence of depression as first episode of bipolar disorder by virtue of earlier age of onset compared to unipolar illness.(11)

Objectives:

The objective of this proposal is to investigate response to acute lithium treatment in subjects who meet the diagnostic criteria for major depression, but are potentially at risk for bipolar disorder, by virtue of family history of bipolarity or completed suicide.

Primary Hypothesis:

Subjects with depression considered at risk for bipolar disorder, will show a significant clinical response to lithium.

Secondary Hypothesis:

1. Subjects with depression considered at risk for bipolar disorder, will show a significant clinical response to paroxetine.
2. Treatment emergent mixed symptoms, in particular agitation, will occur only in the antidepressant treated group.

Study Design:

This is a 6 week double-blind randomized controlled pilot trial of lithium versus paroxetine in subjects with major depression who have either a family history of bipolar disorder or completed suicide. 20 subjects men or women above the age of 18 will be recruited at this centre.

Patients will be randomized to receive either lithium or paroxetine at their first study visit and the dose of drug will be adjusted to find the right one for each patient. Patients will be assessed on a weekly basis thereafter.Data from this pilot study will help in the development of a larger adequately powered study to compare lithium and paroxetine in the treatment of depression in this high risk group.

Patients excluded from the study would include subjects not able to give informed consent,pregnant or breast-feeding women,a current diagnosis of panic disorder, post traumatic stress disorder or psychosis,a history of mania or hypomania,active substance abuse or dependence in the last 6 months, a current depressive episode less than 4 weeks or greater than 12 months in duration, a current or prior adequate trial of lithium or paroxetine,concurrent use of other antidepressants or augmenting agents for the treatment of depression,or a clinically significant medical illness, in particular renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Not currently participating in a drug or medical device clinical trial
* Male or female over the age of 18
* DSM - IV Diagnosis of major depression
* Positive family history of bipolar disorder or completed suicide

Exclusion Criteria:

* Not able to give informed consent
* Pregnant or breast-feeding
* Current additional psychiatric diagnoses including Panic Disorder, Post -Traumatic Stress Disorder (PTSD) or Psychosis
* History of mania or hypomania
* Active substance abuse or dependence in the last 6 months
* Current depressive episode less than 4 weeks or greater than 12 months in duration
* Current or prior adequate trial of lithium or paroxetine
* Current use of other medications such as antidepressants for the treatment of depression
* Clinically significant medical illness, in particular kidney problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Response will be defined as 50% reduction in MADRS score. | weekly
Remission will be defined as MADRS ≤ 12. | weekly
The MADRS will be done at week 0,1,2,3,4,5,6. | weekly

SECONDARY OUTCOMES:
The Hamilton Depression Rating Scale (HAM -D)-17 item scale, at weeks 0 and 6. | weeks 0 and 6
Hamilton Anxiety Rating Scale (HAM-A),at weeks 0 and 6. | weeks 0 and 6
The Young Mania Rating Scale (YMRS), at weeks 0,1,2,3,4,5,6. | weekly
The Bipolar Depression Rating Scale (BDRS) (42),at weeks 0,1,2,3,4,5,6. | weekly
Checklist of DSM IV symptoms of mania/ hypomania, with additional questions assessing the presence of mood lability, abnormally high energy, abnormally high libido, and rage. Done at weeks 0,1,2,3,4,5,6. | weekly
The Beck Suicide Scale (BSS), at weeks 0, 1, 2,3,4,5, 6. | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Claire O'Donovan M O'Donovan, MB FRCPC, Principal Investigator — Capital District Health Authority and Dalhousie University
Locations (1):
- Capital District Health Authority - Dept. of Psychiatry, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Judd LL, Akiskal HS. The prevalence and disability of bipolar spectrum disorders in the US population: re-analysis of the ECA database taking into account subthreshold cases. J Affect Disord. 2003 Jan;73(1-2):123-31. doi: 10.1016/s0165-0327(02)00332-4. PMID 12507745
- [Background] Perugi G, Micheli C, Akiskal HS, Madaro D, Socci C, Quilici C, Musetti L. Polarity of the first episode, clinical characteristics, and course of manic depressive illness: a systematic retrospective investigation of 320 bipolar I patients. Compr Psychiatry. 2000 Jan-Feb;41(1):13-8. doi: 10.1016/s0010-440x(00)90125-1. PMID 10646613
- [Background] Roy-Byrne P, Post RM, Uhde TW, Porcu T, Davis D. The longitudinal course of recurrent affective illness: life chart data from research patients at the NIMH. Acta Psychiatr Scand Suppl. 1985;317:1-34. doi: 10.1111/j.1600-0447.1985.tb10510.x. PMID 3861072
- [Background] Yatham LN, Kennedy SH, O'Donovan C, Parikh S, MacQueen G, McIntyre R, Sharma V, Silverstone P, Alda M, Baruch P, Beaulieu S, Daigneault A, Milev R, Young LT, Ravindran A, Schaffer A, Connolly M, Gorman CP; Canadian Network for Mood and Anxiety Treatments. Canadian Network for Mood and Anxiety Treatments (CANMAT) guidelines for the management of patients with bipolar disorder: consensus and controversies. Bipolar Disord. 2005;7 Suppl 3:5-69. doi: 10.1111/j.1399-5618.2005.00219.x. PMID 15952957
- [Background] Ghaemi SN, Rosenquist KJ, Ko JY, Baldassano CF, Kontos NJ, Baldessarini RJ. Antidepressant treatment in bipolar versus unipolar depression. Am J Psychiatry. 2004 Jan;161(1):163-5. doi: 10.1176/appi.ajp.161.1.163. PMID 14702267
- [Background] Blacker D, Lavori PW, Faraone SV, Tsuang MT. Unipolar relatives in bipolar pedigrees: a search for indicators of underlying bipolarity. Am J Med Genet. 1993 Dec 15;48(4):192-9. doi: 10.1002/ajmg.1320480405. PMID 8135302
- [Background] Bowden CL. A different depression: clinical distinctions between bipolar and unipolar depression. J Affect Disord. 2005 Feb;84(2-3):117-25. doi: 10.1016/S0165-0327(03)00194-0. PMID 15708408
- [Background] Strober M, Carlson G. Bipolar illness in adolescents with major depression: clinical, genetic, and psychopharmacologic predictors in a three- to four-year prospective follow-up investigation. Arch Gen Psychiatry. 1982 May;39(5):549-55. doi: 10.1001/archpsyc.1982.04290050029007. PMID 7092488
- [Background] Hirschfeld RM, Cass AR, Holt DC, Carlson CA. Screening for bipolar disorder in patients treated for depression in a family medicine clinic. J Am Board Fam Pract. 2005 Jul-Aug;18(4):233-9. doi: 10.3122/jabfm.18.4.233. PMID 15994469
- [Background] Koukopoulos A, Faedda G, Proietti R, D'Amico S, de Pisa E, Simonetto C. [Mixed depressive syndrome]. Encephale. 1992 Jan;18 Spec No 1:19-21. French. PMID 1600899
- [Background] Berk M, Dodd S. Are treatment emergent suicidality and decreased response to antidepressants in younger patients due to bipolar disorder being misdiagnosed as unipolar depression? Med Hypotheses. 2005;65(1):39-43. doi: 10.1016/j.mehy.2005.02.010. PMID 15893115